CLINICAL TRIAL: NCT00376545
Title: Brain Connectivity Between Visual Input and Motor Output
Brief Title: Brain Connectivity Between Visual Input and Movement
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060243; 06-N-0243
Record Dates: First submitted 2006-09-14; First posted 2006-09-15 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-11-13

CONDITIONS: Occipital Cortex; Prefrontal Cortex; Healthy
Keywords: Functional Magnetic Resonance Imaging (fMRI); Visuomotor; Occipital Cortex; Prefrontal Cortex; Healthy Volunteer; HV

SUMMARY:
This study will explore how the areas in the brain are connected to link what people see to what they do; that is, how they use what they see to help guide their movements. The study uses functional magnetic resonance imaging (fMRI) to look at different areas in the brain while a person performs tasks in which both what they see (visual input) and what they do (their motor response) are related or unrelated.

Healthy, right-handed normal volunteers who are 18 years of age or older may be eligible for this study. Candidates are screened with a medical history, neurological examination and MRI scan, if one has not been done within a year of entering the study. MRI uses a magnetic field and radio waves to produce images of body tissues and organs. The subject lies on a table that can slide in and out of the scanner (a narrow cylinder), wearing earplugs to muffle loud knocking sounds that occur during scanning. The procedure lasts about 90 minutes, during which the subject is asked to lie still for up to 30 minutes at a time.

Participants undergo fMRI for this 1-day study. fMRI differs from ordinary MRI in that the subject performs tasks during the scanning, allowing researchers to see brain changes that occur during performance of the activity. Before the scan, the subject is trained for the tasks, which include looking at shapes while following them with the fingers and looking at shapes without making finger movements. Following the testing, subjects have a second ordinary MRI scan.

DETAILED DESCRIPTION:
OBJECTIVE:

The purpose is to analyze task-related connectivity changes in brain regions, using a block design blood oxygenation level-dependent functional magnetic resonance imaging (BOLD-fMRI), as a function of the linkage between visual input and motor output.

STUDY POPULATION:

- 25 right-hand dominant, healthy adult volunteers

DESIGN:

Connectivity between brain areas can change related to the dependence level between visual input and motor output. The dependence level will be modulated while performed tasks engage visual and motor areas either in a functionally related fashion or not. Subjects will perform a visuomotor task (VM, dependence level = maximal) that consists of tracking a target by exerting force isometrically on a transducer with their right index finger (target signal and exerted force are displayed in the scanner). In the visual plus motor task (V+M), two different tasks will be performed simultaneously. Subjects will perform the same motor task as in VM but without target signal and visual feedback of their force control, while a neutral visual input unrelated to the motor output is dynamically flashed in the screen. In the visual (V), subjects will watch the target signal while relaxed. In the motor task (M), subjects will produce the same motor task as in VM and V+M while staring at a static fixation cross. A rest period will require subjects to fixate on a stationary dot in the middle of the visual field. fMRI scanning will be used to record brain activity during tasks.

The experimental phase will have six sets of 6-minute scanning sessions where the subject will perform the conditions. The conditions will appear pseudo-randomly throughout the scan sessions. V will always precede VM condition to avoid motor system activation secondary to imagination of movement primed by the visual stimulus. The M and VM conditions will be presented in a random order. At the completion of fMRI scanning, a baseline high-resolution MRI T1 scan will be obtained for anatomic localization and co-registration.

OUTCOME MEASURES:

The primary outcome is the connectivity change in brain networks in response to loss of dependence between a sensory input and the motor output. We will be focused on the correlation between the time series of activations in each condition and the connectivity changes over all the conditions. This will allow us to elucidate the task-dependent connectivity between occipital cortex and prefrontal cortex relative to the functional link between visual input and motor output.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Subjects age 18 and older
* Subjects must be right-hand dominant (Edinburgh Handedness Quotient greater than 60)
* Subjects willing to abstain from caffeine or alcohol for 48 hours prior to the fMRI scanning

EXCLUSION CRITERIA:

* Subjects with any abnormal findings on neurological exam
* Subjects who are pregnant (as determined by a positive urine pregnancy test)
* Subjects with any finding on the MRI safety questionnaire which prevents them from safely undergoing an MRI scan
* Subjects with metallic dental fillings which are likely to cause MRI artifacts
* Subjects with any history of brain tumor, stroke, head trauma or a vascular malformation as obtained by history or from imaging studies
* Subjects with any history of a severe medical condition, such as cardiovascular disease, which would prevent them from lying flat for up to 120 minutes
* Subjects without the capacity to give informed consent
* Subjects with claustrophobia or other restrictions which prevent them from undergoing a scan in a confined space for up to 60 minutes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25
Dates: Start 2006-09-12; Primary Completion 2008-11-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Kaiser J, Lutzenberger W. Human gamma-band activity: a window to cognitive processing. Neuroreport. 2005 Feb 28;16(3):207-11. doi: 10.1097/00001756-200502280-00001. PMID 15706221
- [Background] Singer W, Gray CM. Visual feature integration and the temporal correlation hypothesis. Annu Rev Neurosci. 1995;18:555-86. doi: 10.1146/annurev.ne.18.030195.003011. No abstract available. PMID 7605074
- [Background] von der Malsburg C, Schneider W. A neural cocktail-party processor. Biol Cybern. 1986;54(1):29-40. doi: 10.1007/BF00337113. PMID 3719028